CLINICAL TRIAL: NCT06693921
Title: Artificial Intelligence-Enhanced Three-Dimensional Reconstruction of Combined Horizontal and Vertical Ridge Deficiencies Using Allogenic Dentin Block Versus Shell Tooth Graft Combined With Simultaneous Implant Placement
Brief Title: Artificial Intelligence-Enhanced Three-Dimensional Reconstruction of Ridge Deficiencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant professor of periodontology, faculty of oral and dental medicine, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFSIRB200-312
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Bone Loss
Keywords: deficient ridges; Artifitial intelligence; allograft; ridge reconstruction
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blinded only the outcome assessor is masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- allogenic dentin block (Experimental): Participants will receive allogenic dentin block for reconstruction of combined vertical and horizontal ridge defects with simultaneous implant placement in the maxillary esthetic zone.
  Interventions: Procedure: AI/guided block graft
- allogenic dentin shell (Experimental): Participants will receive allogenic dentin shell for reconstruction of combined vertical and horizontal ridge defects with simultaneous implant placement in the maxillary esthetic zone.
  Interventions: Procedure: AI/guided shell graft

INTERVENTIONS:
Procedure: AI/guided block graft — The allo-dentin tooth graft will be prepared by placing a dentin block from extracted teeth in the trim template and trimming with round burs to the planned dimension under the guidance of the template.
  Arms: allogenic dentin block
Procedure: AI/guided shell graft — The allo-dentin shell graft will be prepared by placing a dentin shell from extracted teeth in the trim template and trimming with round burs to the planned dimension under the guidance of the template
  Arms: allogenic dentin shell

SUMMARY:
n the current study, AI-assisted 3D ridge augmentation of combined vertical and horizontal deficient ridges utilizing allogenic dentin block versus allogenic dentin shell graft will be assessed.

DETAILED DESCRIPTION:
Severe periodontitis, trauma, and long-term edentulism can cause significant resorptive alterations of the alveolar ridge, leading to severe bone defects in the esthetic zone. Careful hard and soft tissue evaluation prior to implant surgery is important to restore proper function and esthetics. Horizontal, vertical, or combined ridge defects after extraction significantly influence dental implant placement and its long-term stability, as well as the final esthetics outcome.

Under natural conditions following a tooth extraction, the alveolar bone around the empty socket would undergo resorption and the alveolar ridge would recede in height and width. Besides leading to aesthetic and functional issues, the reduced bone volume would also cause insufficient support to the dental implant, causing the implant to become loose and unstable. For patients facing such issues, alveolar ridge augmentation is necessary to regenerate the bone tissue and restore the alveolar ridge so as to ensure the long-term stability of the implant.

Although a large number of alloplastic, allogenic or xenogenic bone substitute materials are available for reconstruction of the alveolar crest, the use of autogenous bone is still considered the gold standard. Autogenous bone has excellent osteoinductive, osteoconductive and osteogenetic characteristics; immunological reactions or the transmission of diseases can be safely avoided, and predictable augmentation results can be obtained.

For several years, the use of dentin as an alternative autogenous material for alveolar crest reconstruction and the grafting of bone deficits has been described and investigated in animal experiments and clinical studies. Dentin is a suitable grafting material because it is very similar to bone in its organic and inorganic composition. Similar to the alveolar bone, about 90% of the organic substance of dentin consists of type I collagen. Also, osteogenetically relevant structural proteins, such as osteocalcin, osteonectin, phosphoprotein and sialoprotein, can be found in dentin. Moreover, dentin contains osteogenetically active factors, including bone morphogenetic protein 2 (BMP-2), tissue growth factor-ß (TGF-ß) and insulin- like growth factor-2 (IGF-2). As in alveolar bone, the inorganic components of dentin consist of various calcium phosphates such as hydroxylapatite, ß-tricalcium phosphate, octacalcium phosphate and amorphous calcium phosphate. Compared with autogenous bone, the use of dentin offers the advantage of avoiding the harvesting procedure and the possible resulting donor site morbidity with promising clinical and histological results owing to its inherent osteoinductive and osteoconductive capacity. In comparison to autogenous bone block graft, dentin grafts also show significantly less resorption.

However, autogenous dentin graft has limitations despite its proven bone-formation capacity: dependence of the quantity on the number of teeth indicated for extraction and the condition of the extracted teeth, lack of a standard method to process autogenous dentin graft, and patient preference. Therefore, the application of dentin graft material from other individuals- allogeneic dentin graft-has been considered as an alternative autogenous dentin graft. Allo-dentin graft was conceptualized from the demineralized bone matrix, which was largely developed and defined for the bone induction principle, which states that a protein macromolecule in dentin and bone induces the differentiation of mesenchymal cells into osteoblasts; this was postulated by Urist in 1965. The Allo-dentin graft is a refined allograft that has osteoinductivity and has been clinically used since the 1980s. Very few studies have investigated the application of Allo-dentin graft as bone substitutes for bone graft surgery. The narrative review of revealed that Allo-dentin graft has demonstrated a great potential for osteoinductivity in extraskeletal sites, maximum clinical safety and efficacy without antigenicity nor provoked immunologic reactions.

Cone beam computed tomography (CBCT) imaging developments went hand in hand with the increasing use of 3D imaging applications for presurgical planning and transfer of oral implant treatment. The main reasons for the triumph of CBCT are its capabilities of volumetric jaw bone imaging at reasonable costs and doses, with a relative advantage of having a compact, affordable, and nearby equipment. For the clinicians involved in implant rehabilitation, the power of a dental 3D dataset is not only situated in the diagnostic field, but also in the potential of gathering integrated patient information for presurgical and treatment applications related to oral implant placement. Nowadays, rapid advances of digital technology and computer-aided design/computer-aided manufacturing (CAD/CAM) systems are indeed creating challenging opportunities for diagnosis, surgical implant planning and delivery of implant-supported prostheses.

Segmenting organs and tissues to create 3-dimensional models is a useful technique for diagnosis, surgical planning, and simulation. This technique is also applicable to the planning of 3D-ridge augmentation, which plays a significant part in oral and maxillofacial surgery. Segmentation enables accurate measurement of the ridge volume, providing clinicians with quantitative insight into changes caused by cysts and tumors. In addition, accurately segmenting provides valuable guidance for clinicians when planning ridge augmentation during implant surgery. Although manual segmentation can be used for this purpose, it is time-consuming and dependent on the practitioner's experience due to high inter and intra-observer variability on CBCT images. While artificial intelligence (AI) segmentation is generally more successful and easier to perform than manual segmentation.

In the current study, AI-assisted 3D ridge augmentation of combined vertical and horizontal deficient ridges utilizing allogenic dentin block versus allogenic dentin shell graft will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Insufficient vertical and horizontal bone contour for dental implant placement in the maxillary esthetic zone.

  * Volunteer for participating alveolar bone augmentation by allo-dentin graft technique.
  * Absence of any complicating systemic condition that may contraindicate surgical procedures.
  * Adequate oral hygiene.

Exclusion Criteria:

* Uncontrolled systematic disorders

  * diabetes mellitus
  * uncontrolled periodontal disease
  * history of head and neck radiotherapy
  * pregnancy
  * noncompliant patients
  * uncooperative individuals
  * those unable to attend the study follow-up appointments

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Horizontal buccolingual ridge width | 12 months
  Measuring the buccolingual width of the ridge will be carried out by calculating the distance between the outer boundaries of the palatal and facial bony plates horizontally at a distance 2 mms away from the implant shoulder apically using CBCT.

SECONDARY OUTCOMES:
Facial marginal bone level | 12 months
  Measuring the distance between the fixture shoulder and the facial bone plate crest vertically will be carried out at the fixture midline to determine the facial marginal bone level
Peri-implant bone density | 12 months
  One mm areas of interest were traced 1.2 mm away from the fixture on the CBCT cross-sectional view, followed by counting threshold pixels inside this area to calculate the mean Peri-implant bone density.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kafrelsheikh University, Kafr ash Shaykh
  - Walid Elamrousy, Kafr ash Shaykh

IPD SHARING:
Plan to Share IPD: No
data will not be shared

REFERENCES:
- [Background] Elraee L, Abdel Gaber HK, Elsayed HH, Adel-Khattab D. Autogenous dentin block versus bone block for horizontal alveolar ridge augmentation and staged implant placement: A randomized controlled clinical trial including histologic assessment. Clin Oral Implants Res. 2022 Jul;33(7):723-734. doi: 10.1111/clr.13936. Epub 2022 May 13. PMID 35509125